CLINICAL TRIAL: NCT02969694
Title: Evaluation of Relationship Between Hypersexuality and Psychostimulant Among Men Who Have Sex With Men
Acronym: HYPERCHEM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0746
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psychoactive Substances Consumers
Keywords: addiction; hypersexuality; psychostimulants
MeSH Terms: conditions — Behavior, Addictive; Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who use psychostimulants products in sexual contexts: Patients who come to the CSAPA at the Croix-Rousse Hospital, Lyon France following the use of psychostimulants products in sexual contexts.These patients come for an addictologique support.
  The patients will answer to the G-STAT questionnaire.
  Interventions: Other: G-STAT questionnaire

INTERVENTIONS:
Other: G-STAT questionnaire — Patients will have a consultation with an addiction specialist physician. During the consultation, the physician ask the patient about these sexual practice and the use of psychostimulants. The patient will answer to the G-STAT questionnaire. This questionnaire allows the physician to perform an initial assessment of the patient's sexual addiction.
  The entire consultation takes place in the usual practice of consultations for this addiction.

SUMMARY:
Survey of fifty new psychoactive substances consumers in a context of MTM sexual intercourse.

Evaluation using an hetero-assessment questionnaire about the link between hypersexual disorder and the use of synthetic cathinone.

Evaluation on psychoactive drug addiction, the induced or pre-existing sexual practices and the medico-psycho-social consequences of those practices.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients ≥ 18 years
  * Male homosexual and / or bisexual who come to the CSAPA at the Croix-Rousse Hospital, Lyon France following the use of psychostimulants products in sexual contexts
  * Patients who have received clear information and not opposed to participate in the study
  * Patients affiliated to a social security scheme or similar
  * Patients not undergoing a measure of legal protection
* Exclusion Criteria:

  * Opposition to participation in the study
  * Patients < 18 years
  * Pregnant women or breastfeeding
  * Deprived of individual liberty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who have sex with men and who take psychostimulants products in sexual contexts
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
G-STAT questionnaire | Day 0
  Determine whether there are elements sexual addiction or if its elements are induced by the specific use of psychostimulants. The determination will be made using the interrogation conducted during the CSAPA consultation and G-STAT questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France